CLINICAL TRIAL: NCT06536816
Title: Combined Effects of Game Profile-Based Training and Small-Sided Games on Strength, Endurance, and Performance Among Football Players.
Brief Title: Combined Effects of Game Profile-based Training and Small-sided Games Among Football Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0467
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Physical Endurance; Muscle Strength; Functional Performance
Keywords: Endurance; Strength; Physical Performance

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Game Profile-based training Group (Experimental): 1st group with players having only Game Profile Based training group
  Interventions: Other: Game Profile-based training Group
- Small-sided games Group (Experimental): 2nd group with players having only Small-Sided Games group
  Interventions: Other: Small-sided games Group
- Combined training Group with both Game Profile-based training and Small-sided Games (Experimental): 3rd group with players having both Game Profile-based training and Small-Sided Games group
  Interventions: Other: Combined training Group with both Game Profile-based training and Small-sided Games

INTERVENTIONS:
Other: Game Profile-based training Group — Game profile-based training is a methodology in sports, including football, where training sessions are designed to simulate the specific conditions and challenges that players face during actual games. Coaches analyze individual and team performance data to identify patterns, positions, and scenarios commonly encountered in matches. The training is then structured to replicate these situations, helping players develop the skills, tactics, and decision-making abilities required in real-game scenarios. This approach aims to make training more targeted and relevant to the dynamics of competitive play.
  Arms: Game Profile-based training Group
Other: Small-sided games Group — small-sided game in football, often referred to as a "SSG," is a practice or training activity where players compete in a reduced playing area with fewer players than a full team.
  Arms: Small-sided games Group
Other: Combined training Group with both Game Profile-based training and Small-sided Games — Combined training Group with both Game Profile-based training and Small-sided Games
  Arms: Combined training Group with both Game Profile-based training and Small-sided Games

SUMMARY:
Game profile-based training is a methodology in sports, including football, where training sessions are designed to simulate the specific conditions and challenges that players face during actual games. Coaches analyze individual and team performance data to identify patterns, positions, and scenarios commonly encountered in matches. The training is then structured to replicate these situations, helping players develop the skills, tactics, and decision-making abilities required in real-game scenarios.

DETAILED DESCRIPTION:
This approach aims to make training more targeted and relevant to the dynamics of competitive play, whereas small-sided game in football, often referred to as a "SSG," is a practice or training activity where players compete in a reduced playing area with fewer players than a full team. Small-sided games can vary in size, ranging from 1v1 to 7v7 or 8v8 formats, so integrating game profile-based training with small-sided games creates a comprehensive developmental approach, addressing specific skill needs while providing a dynamic and realistic training environment. This combination can contribute significantly to the overall improvement of football players and the research also involves analyzing the impact of this integrated training methodology on players' technical strength, endurance, and overall performance.

ELIGIBILITY:
Inclusion Criteria:

* Male players
* Age 18-30 years
* Representation of players from various positions
* Players with good health and fitness status
* Participants willing and available for regular assessments
* Athletes playing football with minimum 2-year experience.

Exclusion Criteria:

* Players not actively involved in training and competition
* History of systemic disease
* Prior surgery history
* Participants with irregular attendance or significant deviations from the prescribed training program
* Pre-existing knee pathologies or injuries
* Exclusion of individuals unwilling or unable to participate in regular assessments

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
Endurance | 0 week, 6 weeks, 12 weeks
  The Hoff-test will be used to access endurance among players
Strength | 0 week, 6 weeks, 12 weeks
  The 1 RM test will be used to access strength among players
Performance | 0 week, 6 weeks, 12 weeks
  The Sprint test will be used to access strength among players

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Awais Naeem, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hostrup M, Bangsbo J. Performance Adaptations to Intensified Training in Top-Level Football. Sports Med. 2023 Mar;53(3):577-594. doi: 10.1007/s40279-022-01791-z. Epub 2022 Nov 16. PMID 36380164
- [Background] Bangsbo J. Physiological factors associated with efficiency in high intensity exercise. Sports Med. 1996 Nov;22(5):299-305. doi: 10.2165/00007256-199622050-00003. PMID 8923647
- [Background] Nobari H, Gorouhi A, Mallo J, Lozano D, Prieto-Gonzalez P, Mainer-Pardos E. Variations in cumulative workload and anaerobic power in adolescent elite male football players: associations with biological maturation. BMC Sports Sci Med Rehabil. 2023 Jan 31;15(1):11. doi: 10.1186/s13102-023-00623-5. PMID 36721183
- [Background] da Costa JC, Borges PH, Ramos-Silva LF, Weber VMR, Moreira A, Vaz Ronque ER. Body size, maturation and motor performance in young soccer players: relationship of technical actions in small-sided games. Biol Sport. 2023 Jan;40(1):51-61. doi: 10.5114/biolsport.2023.110749. Epub 2022 Jan 3. PMID 36636197
- [Background] Florez Gil E, Rodriguez-Fernandez A, Vaquera A, Suarez-Iglesias D, Scanlan AT. The discriminative, criterion, and longitudinal validity of small-sided games to assess physical fitness in female basketball players. J Sports Sci. 2023 Sep;41(15):1498-1506. doi: 10.1080/02640414.2023.2279819. Epub 2023 Nov 29. PMID 37947079